CLINICAL TRIAL: NCT03975335
Title: An Intervention Program to Reduce NCD Related Behavioral Risk Factor Among Adolescents in Institutional Settings of Bangladesh
Brief Title: Reducing Behavioral Risk Factors of NCDs: Protocol for a School-based Health Education Program in Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chi Research & Infotec Ltd. (Other)
Collaborators: Directorate General of Health Services (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BSMMU/2018/5958
Record Dates: First submitted 2019-05-14; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Non-communicable Disease Risk Factors
Keywords: NCDs; Risk behaviors; Adolescents; Health education intervention
MeSH Terms: conditions — Risk-Taking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Health education on NCDs and behavioral risk factors was delivered through motivation and observational learning session.
  Interventions: Behavioral: Health education
- Control group (Placebo Comparator): Control group received session on carrier guidance.
  Interventions: Other: Carrier Guidance

INTERVENTIONS:
Behavioral: Health education — In this health education intervention, emphasis is given on evoking adolescents' internal desire to change, supporting self-efficacy to be changed, guiding self-regulatory ways along with facilitating desired changing process by empowering them with choices and skills.
  Arms: Intervention group
Other: Carrier Guidance — Carrier opportunities and counselling
  Arms: Control group

SUMMARY:
This is a before-after designed intervention study conducted in two randomly selected secondary schools- one was selected randomly as intervention school and the another as control school. A baseline survey was conducted among the students of both schools by a pre-tested questionnaire to attain their current status of knowledge, attitude and practices related to NCDs. Afterward, students were enrolled in the intervention group who met the eligibility criteria from the intervention school. The intervention was given through a health promotion session to a group of students, not more than 25 at a time, by trained facilitators. A post-intervention end line survey was conducted among all the participants from both schools using the same questionnaire three months after the baseline survey. An intervention has been developed based on some principals of two psychosocial theory- Motivational Interview and Social Cognitive Theory. Emphasis was given on motivating the adolescents towards a healthy lifestyle, supporting self-efficacy to be changed, guiding self-regulatory ways along with facilitating desired changing process by empowering them with choices about the preventive measures of NCDs. This intervention is expected to increase awareness by equipping the adolescents with specific knowledge and skills and thus, facilitate an eventual change in their practiced risk behaviors.

ELIGIBILITY:
Inclusion Criteria:

• Practicing at least two risk behaviors from three- unhealthy diet, physical inactivity and smoking

Exclusion Criteria:

• Physically disabled or having limited movement

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 823 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Change in knowledge | Three months
  Knowledge about non-communicable diseases related risk behaviors such as dietary habit, physical activity, smoking and alcohol will be measured by 25 knowledge measuring questions scoring 54 in total. Answer to the questions will be regarded as correct or incorrect based on information from standard medical textbooks and guidelines. Difference of knowledge score from pre-intervention to post-intervention survey will be measured.
Change in attitude | Three months
  Attitude towards the risk behaviors- dietary habit, physical activity, smoking and alcohol will be measured by nine attitude measuring questions in a Likert Scale ranging from one to three. Change in attitude score from pre-intervention to post-intervention survey will be measured.
Change in practice | Three months
  Practice will be measured as follows-
  1. Dietary habit: Presence of at least two of the following four habits will be accounted as having dietary risk behavior.
     i. Inadequate fruit consumption: Less than five servings of fruits per day ii. Inadequate vegetable consumption: Less than five servings of vegetables per day iii. Excessive salt consumption: Taking extra or raw salt during every meal iv. Sugar Sweetened Beverage (SSB) consumption: Consuming SSB more than three days per week
  2. Physical activity: Not meeting 60 minutes physical activity of moderate intensity per day will be regarded as physically inactive.
  3. Smoking and alcohol: Smoking regularly in the last 30 days or exposing to passive smoking more than three days per week will be accounted as in risk of smoking. Any amount of alcohol intake or any substance abuse in the last 30 days will be regarded as at risk.
  Change in practice from pre-intervention to post-intervention survey will be measured.

SECONDARY OUTCOMES:
Body Mass Index (BMI) | Three months
  The ratio of body weight in kilogram and the height in meter square will be considered as BMI. Classification of BMI will be done as following- Underweight (Less than 18.5); Normal weight (18.5-24.9); Overweight (25.0-29.9) and Obese (More than 30.0)
Blood Pressure | Three months
  Blood pressure will be measured by an automatic digital sphygmomanometer (HEM-8712, Omron, Kyoto, Japan). Presence of systolic blood pressure ≥ 130 mm of Hg and/or diastolic blood pressure ≥ 80 mm of Hg will be considered as having high blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Md Khalequzzaman, PhD, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh; Sohel Reza Choudhury, DrPH, Study Director — National Heart Foundation Hospital and Research Institute
Locations (1):
- Chi Research & Infotec Ltd., Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No
Study protocol, statistical analysis plan and informed consent form will be shared through

REFERENCES:
- [Derived] Salwa M, Subaita F, Choudhury SR, Khalequzzaman M, Al Mamun MA, Bhuiyan MR, Haque MA. Fruit and vegetables consumption among school-going adolescents: Findings from the baseline survey of an intervention program in a semi-urban area of Dhaka, Bangladesh. PLoS One. 2021 Jun 8;16(6):e0252297. doi: 10.1371/journal.pone.0252297. eCollection 2021. PMID 34101740
- [Derived] Salwa M, Atiqul Haque M, Khalequzzaman M, Al Mamun MA, Bhuiyan MR, Choudhury SR. Towards reducing behavioral risk factors of non-communicable diseases among adolescents: protocol for a school-based health education program in Bangladesh. BMC Public Health. 2019 Jul 25;19(1):1002. doi: 10.1186/s12889-019-7229-8. PMID 31345186